CLINICAL TRIAL: NCT03447925
Title: Treatment of Plantar Keratosis With Medicinal Plant in Diabetic Patients: Randomized, Double-Blind and Controlled Clinical Trial
Brief Title: Treatment of Plantar Keratosis With Medicinal Plant in Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Beatriz Bertolaccini Martínez, Universidade do Vale do Sapucai, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65431417.4.0000.5102
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Keratosis Plantaris
Keywords: callosities; keratosis; diabetes mellitus; plants, medicinal; herbal medicine; keratolytic agents
MeSH Terms: conditions — Callosities; Keratosis; Diabetes Mellitus | interventions — Salicylates; Petrolatum; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicinal Plant X Salicylate (Experimental): Treatment Group (TG) will receive topical treatment with medicinal plant and Salicylate Group (SG) will receive topical treatment with salicylate 10%, both once a day, for 30 consecutive days.
  Interventions: Drug: Medicinal Plant; Drug: Salicylate
- Medicinal Plant X Vaseline (Experimental): Treatment Group (TG) will receive topical treatment with medicinal plant and Control Group (CG) will receive topical treatment with vaseline cream, both once a day, for 30 consecutive days.
  Interventions: Drug: Medicinal Plant; Drug: Vaseline

INTERVENTIONS:
Drug: Medicinal Plant — Medicinal Plant Extract with vaseline cream
  Other Names: Treatment Group (TG)
Drug: Salicylate — Salicylate 10% with vaseline cream
  Other Names: Salicylate Group (SG)
  Arms: Medicinal Plant X Salicylate
Drug: Vaseline — Vaseline cream
  Other Names: Control Group (CG)
  Arms: Medicinal Plant X Vaseline

SUMMARY:
This study evaluates the addition of medicinal plant in the treatment of diabetic foot keratosis. Half of participants will receive medicinal plant and other half will receive a placebo.

DETAILED DESCRIPTION:
Keratosis in feet or plantar callosity is an injury caused by friction or pressure in certain location of the skin. This is a common problem faced by diabetic patients, which usually cause subcutaneous tissue maceration, which favors bacterial invasion. It is responsible for the development of abscesses and ulcers. Ulcer is the main cause of non-traumatic amputation of the feet in diabetic patients. Treatment with medicinal plants is an ancient practice. Brazil has one of the richest floras in the world. Brazilian Ministry of Health recommends the rational use of medicinal plants and encourage the use of this practice by health professionals.

The medicinal plant used in this study is a keratolytic agent, healing, emollient, bactericide and fungicide. The purpose of this study is evaluate the effectiveness of this medicinal plant in the treatment of keratosis in diabetic patients. This study will be controlled, randomized, comparative with standard drug and double-blind. Will be included in the study 90 adult diabetic patients type 1 or 2, with keratosis, both sexes, but do not show feet ulcerated lesions. Patients will be randomised controlled trials in three groups, with 30 people in each, which will receive topical treatment with medicinal plant (treatment group, TG), salicylate 10% (salicylate group, SG) and vaseline cream (control group, CG). The treatment will be once a day, for 30 consecutive days. Numerical scores will be made of the sites with keratosis and individual areas and global measures in the first, 30th days of treatment. The results obtained will be submitted to statistical comparison. This research will follow the standards set by resolution 466/12 of the National Health Council, the Vale do Sapucaí University, for research with human beings and will be conducted in accordance with the ethical recommendations of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

- diabetic patients type 1 and 2 with plantar keratosis

Exclusion Criteria:

- feet ulcerated lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Measures of the sites with plantar keratosis | 30 days
  Measures of the sites with plantar keratosis will be made in the first, and 30th days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beatriz B Martinez, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arosi I, Hiner G, Rajbhandari S. Pathogenesis and Treatment of Callus in the Diabetic Foot. Curr Diabetes Rev. 2016;12(3):179-83. doi: 10.2174/1573399811666150609160219. PMID 26054651
- [Result] Caravaggi C, Sganzaroli A, Galenda P, Bassetti M, Ferraresi R, Gabrielli L. The management of the infected diabetic foot. Curr Diabetes Rev. 2013 Jan 1;9(1):7-24. PMID 22934545